CLINICAL TRIAL: NCT01198938
Title: Postoperative Melatonin Administration and Delirium Prevention in Patients Undergoing Vascular and Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UHN090334B
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery, delirium, melatonin
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melatonin (Active Comparator)
  Interventions: Other: Melatonin

INTERVENTIONS:
Other: Melatonin — Melatonin 5 mg sublingually given at 9 p.m. for 5 postoperative days or until discharge

SUMMARY:
The investigators plan to evaluate the effect of postoperative melatonin administration on postoperative delirium in patients undergoing vascular and cardiac surgery. A total of 302 patients older than 60, undergoing elective vascular surgery will be randomly divided into 2 groups: treatment and control. During the first 5 postoperative days patients will receive sublingually either melatonin 5 mg or placebo at 9:00 pm. The patients will be assessed for the signs of delirium, quality of sleep and severity of pain daily for the first postoperative week. Screening of delirium will be performed by the specially trained research assistant and based on the Confusion Assessment Method and the validated chart review. Diagnosis of delirium will be confirmed by the psychiatrist. Incidence of delirium will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent vascular surgery, with an expected length of stay ≥ 48hours, ASA categories I to IV, signed informed consent, age >60

Exclusion Criteria:

* Lack of informed consent, ASA category V, history of psychiatric illness (schizophrenia, psychosis, bipolar disorder, major depression), Mini Mental State Examination score (MMSE) ≤ 24, history of autoimmune disease, liver cirrhosis, minimally invasive procedures (endovascular aneurysm repair ), history of chronic insomnia, chronic benzodiazepines and/or hypnotics use ( > 3 times /week during a month prior to surgery), treatment with tricyclic antidepressants within a month prior to surgery, history of seizures, allergy to placebo ingredients or melatonin ( WN Pharmaceuticals.LTD), melatonin consumption in the last months prior to surgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | preoperative assessment up to 7 days postoperatively

SECONDARY OUTCOMES:
Pain score, using the standard 10-cm visual analog score (0-no pain, 10-worst, unbearable pain) | Preoperative assessment upt to 7 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital, UHn
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada